CLINICAL TRIAL: NCT06359093
Title: Prevalence Of Non-Carious Cervical Lesions, Associated Risk Indicators and Salivary Assessment Among Middle Adulthood Patients Attending the Cairo University Dental Educational Hospital: Analytical Cross-Sectional Study
Brief Title: Prevalence Of Non-Carious Cervical Lesions, Associated Risk Indicators and Salivary Assessment Among Middle Adulthood Patients.
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rowayda Anwar Hosny Eltarawy, Assistant Lecturer, Cairo University
Other Study IDs: 14422023557605
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Non-carious Cervical Lesions
Keywords: patient-related risk factors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to describe the prevalence of non-carious cervical lesions in middle adulthood patients attending the Cairo University Dental Educational Hospital and to analyze the distribution of lesions by gender and age, tooth functional group, jaw, arch side and tooth surface. Moreover, to explore the associated risk indicators of the lesions as well as the flow rate and pH of saliva, as one of the potential etiological factors, will be assessed.

DETAILED DESCRIPTION:
Dental patients will be recruited from diagnostic central clinic at the Cairo University Dental Educational Hospital. Oral examination will be done, the full aim of the study will be explained to the patient, and patient acceptance is a must. The questionnaire will be filled by patients including age, gender, occupation, education, place of residence, toothbrushing: included frequency, method, intensity, hardness and duration, biting and chewing habits, medical history [related to gastrointestinal problems such as belching, heartburn, vomiting, gastro-oesophageal reflux (GER), peptic ulcer disease], eating disorders (anorexia, bulimia), medication list, frequency of consuming acidic food and fruits, carbonated beverages and alcohol and smoking status. Salivary assessment regarding flow rate and pH for a subgroup diagnosed with non-carious cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age between 41-60 years old.
2. Patient consulting in the outpatient clinic
3. Provide informed consent.
4. Males & Females
5. Egyptian

Exclusion Criteria:

1. Patients under or over this age group.
2. Refuse to participate in the study.
3. Wearing orthodontic appliance.
4. The presence of trismus.

Ages: 41 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Middle adulthood patients (41-60 years old) attending Diagnostic central clinic at the Cairo University Dental Educational Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1532 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of non-carious cervical lesions (NCCLs) in Middle adulthood patients (41-60 years old) attending Diagnostic central clinic at the Cairo University Dental Educational Hospital. | Day 1
  clinical examination

SECONDARY OUTCOMES:
Associated risk indicators for all participants. 3.Salivary assessment regarding flow rate and pH for subgroup diagnosed with non-carious cervical lesions. | Day 1
  questionnaire will be used to collect data. For quantitative analysis of saliva: if saliva flow rate is less than 1ml/min , it is considered xerostomia.
  If saliva flow rate is less than 1ml/min , it is low salivary flow if saliva flow rate is more than 3, it is high salivary flow

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt